CLINICAL TRIAL: NCT05004259
Title: The Safety of Repurposing Daratumumab for Relapsed or Refractory Autoimmune Antibody Mediated Hemolytic Anemia
Acronym: DARA-AIHA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Matthew R. Sullivan, Assistant Professor of Medicine, Geisel School of Medicine, Dartmouth, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY02000992 21SUL992
Record Dates: First submitted 2021-07-28; First posted 2021-08-13 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-01

CONDITIONS: Hemolytic Anemia
MeSH Terms: conditions — Anemia, Hemolytic | interventions — daratumumab; Hyaluronoglucosaminidase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm 1 (Experimental): Six weekly doses of subcutaneous daratumumab 1,800mg and hyaluronidase 30,000U.
  Interventions: Drug: Daratumumab / Hyaluronidase Injection

INTERVENTIONS:
Drug: Daratumumab / Hyaluronidase Injection — Subcutaneous injection of daratumumab and hyaluronidase

SUMMARY:
A single-arm study utilizing a 6 x 4 expansion design using daratumumab SC treatment for patients with refractory Autoimmune Hemolytic Anemia.

DETAILED DESCRIPTION:
Autoimmune Hemolytic Anemia (AIHA) is a hematologic disorder in which the red blood cells are targeted and destroyed by autoantibodies produced by the immune system, specifically B-cells and plasma cells. It can be either idiopathic, or secondary to other autoimmune conditions, but is commonly related to lymphoproliferative disorders such as CLL or indolent lymphomas. It is a rather uncommon condition, which affects an estimated 17 people per 100,000 in their lifetime.

Unfortunately, AIHA is often difficult to treat. The goal of treatment is to achieve and maintain a Hemoglobin concentration of above 10 g/dL. Treatment historically involves the use of relatively high doses of steroids (i.e. 1 mg/kg), followed by a prolonged taper. According to a review article, 80% of patients initially respond to corticosteroid therapy, but steroids alone do not frequently "cure" the disorder, as steroids do not eliminate the anti-RBC antibody producing clone. In fact, only 20% of patients treated with first line steroid therapy are cured, and 15-20% of patients require maintenance Prednisone doses above 15 mg per day. This puts patients at risk of long-term steroid side effects, including infections, osteoporosis, aseptic joint necrosis, diabetes and hypertension.

The discovery of rituximab improved outcomes for AIHA. Rituximab is a monoclonal antibody against CD20, a marker for B-cells, that is now approved in both the first-line setting as well as relapsed/ refractory AIHA. It works by depleting CD20-positive B-cells that produce the autoantibody.

Early studies have shown that adding rituximab to steroids as first line treatment improved outcomes compared to steroids alone. In one study, a similar number of patients responded to rituximab and steroid, compared to steroid alone, but the length of response was significantly improved for the rituximab arm. Among responders, at 36 months, 70% vs 45% of patients treated in the combination arm vs steroids alone were still in remission.

However, despite these advances, some patients either fail to respond to the rituximab (20-30%), or have to remain on unacceptably high doses of steroid to control their hemolysis. In addition, many relapse after rituximab therapy. At that point, splenectomy is commonly recommended, but this only has a cure rate of 20%, is invasive, and comes with long-term sequelae of risks of clots and infection. After splenectomy, patients are left with a host of other immunosuppressants, such as azathioprine, mycophenolate, cyclosporine, or cyclophosphamide, but these typically require long term usage, and have poor side effect profiles (infection, liver toxicity, renal toxicity, lymphoma, etc), and are often ineffective.

Given the need for therapeutic options for patients with refractory or relapsed AIHA who have already received treatment with steroids and rituximab, this study proposes use of daratumumab therapy in this patient population. Daratumumab is a CD38-directed cytolytic monoclonal antibody and is approved for use in patients with multiple myeloma. CD38 is an attractive target in AIHA, because it is expressed not only on B-cells, but also on plasma cells, which rituximab does not target (see figure below for the evolution of CD markers in B-cell maturation). CD38+ plasma cells may be an important source of resistance to rituximab, as they can survive a long time and continue to produce the anti- red blood cell (RBC) antibodies.

In support of the investigator hypothesis, a case report study of three post-allogeneic transplant patients with AIHA refractory to steroids, rituximab, and proteosome inhibition, treated with daratumumab indicated promising results. Two out of the three patients were cured while the third patient had a transient response and relapsed eight months later. Similar results have been reported by other institutions, again in case report form. In addition, daratumumab has also been successfully utilized for refractory Immune Thrombocytopenia (ITP) in the post-transplant setting.

Additionally, here at Dartmouth clinicians have a short history of off labeled use in a 20 year old male with refractory Evans Syndrome, involving AIHA, ITP, and autoimmune neutropenia. Over the years, he had received multiple lines of immunosuppressant agents, but he was refractory to or relapsed quickly after all treatments. Based on the above literature, the Hematology team tried daratumumab, which produced a dramatic improvement in all cell lines within 2 weeks. He was then transferred to the National Institute of Health, where he received an allogeneic stem cell transplant, which would not have been possible without first gaining control over his autoimmune cytopenias with the use of daratumumab therapy.

The investigators of this trial have found daratumumab SC to be safe and very tolerable in the treatment of Multiple Myeloma. Given the strong scientific rationale to support the use of daratumumab in treating patients with relapsed/refractory AIHA, this trial aims to study the safety of daratumumab in this new patient population. The investigators expect to demonstrate safety of daratumumab treatment in patients with AIHA, and to observe clinical response, which will support future larger-scale clinical trials.

As mentioned previously, daratumumab SC has been studied and approved in multiple myeloma and light chain amyloidosis. Of note, the literature reports different pharmacokinetics in each disease; this is thought to perhaps be reflective of a varying burden of plasma cells between the diseases. The half-life associated with the linear clearance of daratumumab is 20 days in patients with multiple myeloma and 28 days in patients with light chain amyloidosis, according to the Darsalex Faspro product label. The pharmacokinetics of daratumumab in patients with relapsed/refractory AIHA is unknown and may differ from other indications where daratumumab is used. To study this, the investigators will measure daratumumab levels at baseline, weekly before treatments, and then at time points 14 and 28 days after the last dose. The serum Cmin (Ctrough) concentrations of daratumumb will be measured in the Clinical Pharmacology Shared Resource using the commercially available the ELISA assay (Eagle Biosciences). Appropriate modeling using WinNonLn pharmacokinetic-pharmacodynamic (PK-PD) software will be used to determine primary pharmacokinetic parameter and explore PK-PD using non-linear models such as the Sigmoid Emax model.

Also, because the investigator hypothesis is based on the investigator expectation that daratumumab will kill the plasma cells responsible for producing the anti-RBC antibodies, the investigators will also measure the anti-RBC antibody levels at baseline, at week 6 of treatment, and then at 3 months after the last dose; RBC antibody levels will be compared to clinical response to evaluate potential correlation. The investigators do appreciate that daratumumab does bind to RBCs via low expression of CD38 on RBCs. However, the Dartmouth-Hitchcock Medical Center Blood Bank Director believes that by pretreating the test cells to remove CD38, the investigators can effectively remove the daratumumab from the specimen, and therefore proceed to use dilutional methods to quantify the anti-RBC level.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have confirmed autoimmune hemolytic anemia, based on a Hemoglobin <10 g/dL, a positive Direct Antiglobulin Test, elevated LDH, and elevated Reticulocyte count, low Haptoglobin test.
* Patients must have been previously treated with both a course of steroids starting at a dose of at least 1mg/kg of Prednisone (or steroid equivalent) and at least 100mg of rituximab previously. They must show signs of ongoing hemolysis (as above) either 1) recurring after previous treatment, 2) or while on a Prednisone dose (or equivalent) of 10mg daily or greater.
* Age ≥18 years
* Patients are allowed to be on steroids, as per standard of care. The dosing regimens may include up to 1mg/kg of Prednisone followed by a Prednisone taper, or a regimen of 40mg of Dexamathasone for 4 days. (See Section 6.13 for recommended steroid taper.)
* All patients must give informed consent indicating they are aware of the investigational nature of this treatment, as well as the study protocols and requirements.
* Patients with Evan's syndrome are permissible
* Patients must have performance status of ECOG 0-2

Exclusion Criteria:

* Patients with active HIV, Hepatitis B, Hepatitis C. We define active as having a detectable viral load. Patients with a prior exposure or well controlled disease while on treatment will be permitted. More information regarding management of these infections can be found in the footnote of the schema in Section 6.1.
* Patients with active Systemic Lupus Erythematosus with other systemic organ involvement requiring treatment
* Patients with active lymphoid malignancy, other than Chronic Lymphoid Leukemia or other low grade lymphoproliferative disorders, not otherwise requiring treatment. Patients with a history of solid tumors are allowed, but must not have received treatment (chemotherapy, surgery, etc.) for a malignancy within 3 years before the date of randomization (exceptions are squamous and basal cell carcinomas of the skin, carcinoma in situ of the cervix or breast, or other non-invasive lesion), which is considered cured with minimal risk of recurrence within 3 years.
* Patients with a serious uncontrolled medical disorder or active infection which would impair their ability to receive study treatment will be excluded. Significant cardiac disease, including uncontrolled high blood pressure, unstable angina, congestive heart failure, myocardial infarction within the previous 3 months or serious cardiac arrhythmias will be excluded. Dementia or significantly altered mental status that would prohibit the understanding or rendering of informed consent and compliance with the requirements of this protocol will be excluded.
* Patients who are pregnant or breastfeeding
* COPD with an FEV1 <50% predicted, or moderate or severe persistent asthma within the past 2 years, or uncontrolled asthma of any classification
* Renal failure with GFR <20 ml/min
* End stage liver disease, as defined by local guidelinesEnd stage liver disease, as defined by local guidelines
* Prior treatment with daratumumab or any other anti-CD38 therapies
* Exposure to an investigational drug (including investigational vaccine) or invasive investigational medical device for any indication within 4 weeks or 5 pharmacokinetic half-lives, whichever is longer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2024-09-21 (Actual); Study Completion 2024-09-21 (Actual)

PRIMARY OUTCOMES:
Determine safety of treatment | Up to 10 weeks
  Monitor for safety by cataloging any infections, injection site reactions or systemic reactions and any other adverse events that occur during the study period. The investigator will also catalog all adverse events, to monitor for any unpredicted side effects in this new patient population, as judged by the treating provider.
Determine dose-limiting toxicities | Up to 6 weeks
  Using a 6 by 4 expansion design in which the study will be stopped if a subject experiences unacceptable toxicity. Unacceptable toxicity is defined as 2 of the first 6 patients experiencing either: Grade 3 or higher infection of any organ system or Grade 3 or higher systemic reactions

SECONDARY OUTCOMES:
Determine the overall response rate (ORR) of daratumumab in patients with relapsed/refractory AIHA | Up to 18 weeks
  Assess the percentage of patients who achieve a complete response (CR) or a partial response (PR). CR is determined by the normalization of hemoglobin concentration without immunosuppressive treatment or steroids and no evidence of active hemolytic activity. PR is defined as increase in hemoglobin to above 10 g/dL without transfusions, having evidence of ongoing hemolysis based on elevated LDH and/or reticulocyte count and/or bilirubin level, and requiring low-dose steroid (less than or equal to 10mg/day or steroid equivalent) to maintain hemoglobin level greater than 10 g/dL.
Determine the time to next treatment (TTNT) | Through study completion, an average of 1 year
  TTNT is defined as the time the time in months from the first dose of daratumumab until the time to a new treatment.

OTHER OUTCOMES:
Trough Plasma Concentration (Cmin) | Pre-treatment through 28 days after the last dose of study treatment
  Measure daratumumab trough levels at baseline, during treatment, and days 14 and 28 post -last dose. The serum Cmin (Ctrough) consentrations of the daratumumab will be measured using the ELISA assay. Appropriate modeling using WinNonLn pharmacokinetic-pharmacodynamic software will be used to determin primary pharmacokinetic parameter and explore pharmacokinetic-pharmacodynamic using non-linear models such as the Sigmoid Emax model.
Assess the change or elimination of anti-Red Blood Cell (RBC) antibody production | Up to 6 weeks
  Cells from blood collection will be pretreated to remove CD38, using an established dithiothreitol (DTT)-based method that has been validated to resolve the daratumumab interference with blood compatibility testing, before diluting the sample to titer the anti-RBC antibody level.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Sullivan, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eaton WW, Rose NR, Kalaydjian A, Pedersen MG, Mortensen PB. Epidemiology of autoimmune diseases in Denmark. J Autoimmun. 2007 Aug;29(1):1-9. doi: 10.1016/j.jaut.2007.05.002. Epub 2007 Jun 19. PMID 17582741
- [Background] Lechner K, Jager U. How I treat autoimmune hemolytic anemias in adults. Blood. 2010 Sep 16;116(11):1831-8. doi: 10.1182/blood-2010-03-259325. Epub 2010 Jun 14. PMID 20548093
- [Background] Birgens H, Frederiksen H, Hasselbalch HC, Rasmussen IH, Nielsen OJ, Kjeldsen L, Larsen H, Mourits-Andersen T, Plesner T, Ronnov-Jessen D, Vestergaard H, Klausen TW, Schollkopf C. A phase III randomized trial comparing glucocorticoid monotherapy versus glucocorticoid and rituximab in patients with autoimmune haemolytic anaemia. Br J Haematol. 2013 Nov;163(3):393-9. doi: 10.1111/bjh.12541. Epub 2013 Aug 24. PMID 23981017
- [Background] Reynaud Q, Durieu I, Dutertre M, Ledochowski S, Durupt S, Michallet AS, Vital-Durand D, Lega JC. Efficacy and safety of rituximab in auto-immune hemolytic anemia: A meta-analysis of 21 studies. Autoimmun Rev. 2015 Apr;14(4):304-13. doi: 10.1016/j.autrev.2014.11.014. Epub 2014 Dec 9. PMID 25497766
- [Background] Zanella A, Barcellini W. Treatment of autoimmune hemolytic anemias. Haematologica. 2014 Oct;99(10):1547-54. doi: 10.3324/haematol.2014.114561. PMID 25271314
- [Background] Schuetz C, Hoenig M, Moshous D, Weinstock C, Castelle M, Bendavid M, Shimano K, Tolbert V, Schulz AS, Dvorak CC. Daratumumab in life-threatening autoimmune hemolytic anemia following hematopoietic stem cell transplantation. Blood Adv. 2018 Oct 9;2(19):2550-2553. doi: 10.1182/bloodadvances.2018020883. PMID 30291113
- [Background] Even-Or E, Naser Eddin A, Shadur B, Dinur Schejter Y, Najajreh M, Zelig O, Zaidman I, Stepensky P. Successful treatment with daratumumab for post-HSCT refractory hemolytic anemia. Pediatr Blood Cancer. 2020 Jan;67(1):e28010. doi: 10.1002/pbc.28010. Epub 2019 Sep 22. PMID 31544339
- [Background] Tolbert, Vanessa P., et al.
- [Background] Migdady Y, Ediriwickrema A, Jackson RP, Kadi W, Gupta R, Socola F, Arai S, Martin BA. Successful treatment of thrombocytopenia with daratumumab after allogeneic transplant: a case report and literature review. Blood Adv. 2020 Mar 10;4(5):815-818. doi: 10.1182/bloodadvances.2019001215. PMID 32119735
- [Background] Blennerhassett R, Sudini L, Gottlieb D, Bhattacharyya A. Post-allogeneic transplant Evans syndrome successfully treated with daratumumab. Br J Haematol. 2019 Oct;187(2):e48-e51. doi: 10.1111/bjh.16171. Epub 2019 Aug 23. No abstract available. PMID 31441030
- [Background] Hill QA, Hill A, Berentsen S. Defining autoimmune hemolytic anemia: a systematic review of the terminology used for diagnosis and treatment. Blood Adv. 2019 Jun 25;3(12):1897-1906. doi: 10.1182/bloodadvances.2019000036. PMID 31235526
- [Background] Chapuy CI, Aguad MD, Nicholson RT, AuBuchon JP, Cohn CS, Delaney M, Fung MK, Unger M, Doshi P, Murphy MF, Dumont LJ, Kaufman RM; DARA-DTT Study Group* for the BEST Collaborative. International validation of a dithiothreitol (DTT)-based method to resolve the daratumumab interference with blood compatibility testing. Transfusion. 2016 Dec;56(12):2964-2972. doi: 10.1111/trf.13789. Epub 2016 Sep 7. PMID 27600566
- [Background] Go RS, Winters JL, Kay NE. How I treat autoimmune hemolytic anemia. Blood. 2017 Jun 1;129(22):2971-2979. doi: 10.1182/blood-2016-11-693689. Epub 2017 Mar 30. PMID 28360039